CLINICAL TRIAL: NCT05988879
Title: A Clinical Research on Functional Cure Strategies for Hepatitis B Among HIV/HBV Co-infected Patients in China
Brief Title: Functional Cure of Hepatitis B in HIV/HBV Co-infected Patients
Status: Recruiting | Type: Observational
Sponsor: Guangzhou 8th People's Hospital (Other)
Responsible Party: Principal Investigator, Linghua LI, Chief physician, Guangzhou 8th People's Hospital
Other Study IDs: GZ8H-202316253
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: AIDS; Hepatitis B
Keywords: HIV/HBV co-infection; Functional cure; Interferon
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis B | interventions — peginterferon alfa-2b

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During the study, the blood sample of patients should be preserved to detect the HIV RNA load , HBV DNA load and ; other co-infected microbes and drug toxicity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ART combined with interferon group: The treatment protocol is ART combined with pegylated interferon α-2b injection. The pegylated interferon α-2b injection is administered subcutaneously at a dose of 180ug once a week. Follow-up times are at baseline, and during treatment at weeks 4, 8, 12, 24, 36, 48, 60, and 72.
  Interventions: Drug: Peginterferon alfa-2b Injection
- ART group: Continuously using ART treatment, without the use of interferon. Follow-up times are at baseline, and during treatment at weeks 12, 24, 36, 48, 60, and 72.

INTERVENTIONS:
Drug: Peginterferon alfa-2b Injection — The pegylated interferon α-2b injection is administered subcutaneously at a dose of 180ug once a week.
  Groups: ART combined with interferon group

SUMMARY:
Evaluate the potential of ART combined with interferon therapy to achieve functional cure of hepatitis B in HIV/HBV co-infected patients

DETAILED DESCRIPTION:
This is a prospective, non-randomized, clinical observational cohort study. The subjects are the advantageous population for functional cure of hepatitis B in HIV/HBV co-infected patients . Depending on whether interferon therapy is used in the real world , the patients are divided into two groups: the ART combined with interferon group and the ART alone group, with 30 cases in each group. Hepatitis B surface antigen seroclearance rate and seroconversion rate will be observed during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old, gender unrestricted.
2. Meeting the People's Republic of China Health Industry Standard (WS293-2008) - "AIDS and HIV Infection Diagnostic Criteria", confirmed as HIV-1 infected.
3. HBsAg positive for more than 6 months.
4. At least 1 year of ART treatment prior to screening, and currently undergoing ART treatment with HBsAg <1000IU/mL, HBeAg negative, HBV DNA <100IU/ml, CD4+T lymphocyte count >200 cells/μL and HIV-RNA<20 copies/ml.

Exclusion Criteria:

1. Pregnant, nursing, planning pregnancy, or with severe mental disorders or uncontrolled epilepsy.
2. Co-infected with Hepatitis A, C, D, or E viruses.
3. With other chronic liver diseases like autoimmune hepatitis, drug-induced hepatitis, alcoholic hepatitis, genetic metabolic liver diseases, or moderate to severe fatty liver.
4. With autoimmune diseases like rheumatoid arthritis, psoriasis, or lupus.
5. Post organ transplant, planning organ transplant, diagnosed or suspected of liver cancer or other malignant tumors, or undergoing immunosuppressive treatment.
6. With severe diseases of heart, lungs, kidneys, brain, retinal disorders, or uncontrolled hypertension or diabetes.
7. Excessive alcohol (average daily alcohol intake >40g for men, >20g for women) or drug users.
8. Participated in other interventional trials within the last three months, or other situations deemed inappropriate for inclusion by researchers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All study participants come from the HIV/HBV co-infection cohort at the Guangzhou Eighth People's Hospital.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2026-08-02 (Estimated); Study Completion 2028-08-02 (Estimated)

PRIMARY OUTCOMES:
Hepatitis B surface antigen seroclearance | 48 weeks
  Hepatitis B surface antigen quantification less than 0.05 IU/mL.

SECONDARY OUTCOMES:
Hepatitis B surface antigen seroconversion | 48 weeks
  Clearance of surface antigen concurrently accompanied by the production of surface antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Linghua Li, PhD, Study Chair — Guangzhou Eighth People's Hospital
Locations (1):
- Guangzhou Eighth People's Hospital, Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No